CLINICAL TRIAL: NCT06122857
Title: Trends of Cancer Incidence and Mortality in Russia: the Breakpoint and Age-period-cohort Analyses of Cancer Incidence and Mortality
Brief Title: Trends of Cancer Incidence and Mortality in Russia
Status: Active, not recruiting | Type: Observational
Sponsor: ITMO University (Other)
Responsible Party: Sponsor
Other Study IDs: FSER-2022-0013
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Oncology; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to assess the dynamics of incidence and mortality for all major groups of cancers for which the national data is available for the longest possible time series. The data obtained from publicly available sources are used.

ELIGIBILITY:
Non applicable

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patient population, that were diagnosed and registered in regions covered by PBCR.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Cancer incidence | 30 years
Cancer mortality | 30 years

CONTACTS AND LOCATIONS:
Locations (1):
- ITMO University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided